CLINICAL TRIAL: NCT02881099
Title: Parkinson's Repository of Biosamples and Network Datasets (Tracking Parkinson's)
Acronym: PRoBaND
Status: Completed | Type: Observational
Sponsor: South Glasgow University Hospitals NHS Trust (Other)
Collaborators: Parkinson's UK (Other); University of Bristol (Other); Cardiff University (Other); University of Glasgow (Other)
Responsible Party: Principal Investigator, Dr Donald Grosset, Senior Research Fellow, University of Glasgow
Other Study IDs: GN11NE062
Record Dates: First submitted 2013-02-01; First posted 2016-08-26 (Estimated); Last update posted 2024-11-29 (Actual); Status verified 2024-11

CONDITIONS: Parkinson's Disease
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — DNA and -80 degrees Centrigrade frozen serum samples
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (3):
- Recent diagnosis (P3): Primary cohort; participants recruited if diagnosed within the last three years
- Early diagnosis (P50): Participants recruited if diagnosed before the age of 50 years old
- Relatives (R): Siblings of existing participants

SUMMARY:
Prospective observational study of Parkinson's disease with repeat clinical assessment and biobanking of blood samples.

DETAILED DESCRIPTION:
To identify genetic and biomarker factors which affect the expression of Parkinson's Disease.

Primary objective: To define the severity and rates of progression of clinical features of Parkinson's Disease.

Secondary objective: To relate clinical phenomenology of Parkinson's disease to genetic and biomarker changes.

ELIGIBILITY:
A. Parkinson's Disease patients

Inclusion criteria

1. Diagnosis of Parkinson's disease, based on UK Brain Bank criteria and made within the preceding 3 years ('recent onset cases') or diagnosed at under 50 years ('under 50 years cases')
2. Age ≥18 to <90years
3. Subject is able and willing to provided informed consent.

Exclusion criteria

1. Patient has severe comorbid illness that would prevent full study participation
2. Patient has features indicating another type of degenerative parkinsonism, e.g. progressive supranuclear palsy
3. Drug-induced parkinsonism (Drug-unmasked PD is allowed)
4. Symmetrical lower body parkinsonism attributable to significant cortical and/or subcortical cerebrovascular disease (patients with 'incidental' small vessel disease on brain imaging are allowed).
5. Negative or normal functional imaging of the presynaptic dopamine system
6. The presence of UK Brain Bank exclusion criteria will be recorded at baseline, allowing for the presence of 1 or 2 exclusion criteria (e.g. dopamine antagonist Drug used; more than one affected relative) (if justified e.g. by abnormal SPECT).

B. First degree relatives Inclusion criteria

1. Age ≥18 to < 90years
2. Resident in the United Kingdom and able to access one of the PRoBaND study centres.
3. Subject is able and willing to provided informed consent.

Exclusion criteria

1. Subject has severe comorbid illness that would prevent study participation
2. Subject already has a diagnosis of Parkinson's disease

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Parkinson's Disease defined by UK Brain Bank criteria Siblings of cases of Parkinson's disease
Sampling Method: Non-Probability Sample
Enrollment: 2614 (Actual)
Dates: Start 2011-11-13 (Actual); Primary Completion 2022-12-31 (Actual); Study Completion 2022-12-31 (Actual)

PRIMARY OUTCOMES:
Proportion of participants with Parkinson's who have gene mutations and variations | Up to 36 months
  Genotyping for leucine rich repeat kinase 2 (LRRK2), Glucocerebrosidase (GBA) (all cases) and Parkin, Phosphatase and tensin homolog-induced putative kinase 1 (PINK1)(onset<50years)

SECONDARY OUTCOMES:
Categorisation of subtypes of Parkinson's using cluster analysis | At 4 years
  Clustering of motor and non-motor features measured using Movement Disorder Society Unified Parkinson's disease rating scale (MDS-UPDRS), Montréal cognitive assessment (MoCA), Non-motor symptom Scale (NMSS), Scale for outcomes in Parkinson's autonomic (SCOPA-AUT), Olfaction testing using University of Pennsylvania Smell Identification Test (UPSIT) or Sniffin' sticks, and Leeds anxiety and depression scale (LADS).
  This will use sequential factor analysis of the results of the above assessments, followed established methods, firstly exploratory factor analysis and secondly confirmatory factor analysis. Factor scores and other clinically important variables will then be combined to construct a single dataset for carrying out the cluster analysis. Hierarchical clustering will then be applied, and models with between 2 and 5 clusters will be described and compared.
Proportion of cases with Parkinson's who have vascular comorbidity and risk factors | At 4 years
  Prior history of vascular events, or calculated using Quantification of Risk version 2 (QRISK2) vascular risk score

CONTACTS AND LOCATIONS:
Overall Officials: Donald Grosset, BSc, MD, Study Director — University of Glasgow

IPD SHARING:
Plan to Share IPD: Yes
Data sharing will be managed to Data & Biosample Access Committee and through direct partnerships with organisations.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Data & Biosample Access manage applications for access for the duration of the grant until 31 December 2023, after which point data will be accessible to researchers through other bodies, including Critical Path for Parkinson's and Global Parkinson's Genetics Program.
Access Criteria: https://c-path.org/programs/cpp/ https://gp2.org/
URL: https://www.trackingparkinsons.org.uk/

REFERENCES:
- [Derived] Malek N, Weil RS, Bresner C, Lawton MA, Grosset KA, Tan M, Bajaj N, Barker RA, Burn DJ, Foltynie T, Hardy J, Wood NW, Ben-Shlomo Y, Williams NW, Grosset DG, Morris HR; PRoBaND clinical consortium. Features of GBA-associated Parkinson's disease at presentation in the UK Tracking Parkinson's study. J Neurol Neurosurg Psychiatry. 2018 Jul;89(7):702-709. doi: 10.1136/jnnp-2017-317348. Epub 2018 Jan 29. PMID 29378790
- [Derived] Swallow DM, Lawton MA, Grosset KA, Malek N, Klein J, Baig F, Ruffmann C, Bajaj NP, Barker RA, Ben-Shlomo Y, Burn DJ, Foltynie T, Morris HR, Williams N, Wood NW, Hu MT, Grosset DG. Statins are underused in recent-onset Parkinson's disease with increased vascular risk: findings from the UK Tracking Parkinson's and Oxford Parkinson's Disease Centre (OPDC) discovery cohorts. J Neurol Neurosurg Psychiatry. 2016 Nov;87(11):1183-1190. doi: 10.1136/jnnp-2016-313642. Epub 2016 Sep 26. PMID 27671901